CLINICAL TRIAL: NCT02849301
Title: Cervical Pessary in Women With Arrested Preterm Labor and Short Cervix
Acronym: PWK
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: different protocol started, new registration
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Gabriele Saccone, MD, Federico II University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2378
Record Dates: First submitted 2016-07-27; First posted 2016-07-29 (Estimated); Last update posted 2018-11-19 (Actual); Status verified 2018-11

CONDITIONS: Preterm Birth
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cervical pessary (Experimental): Arabin cervical pessary
  Interventions: Device: Arabin cervical pessary
- Standard care (No Intervention): No treatment

INTERVENTIONS:
Device: Arabin cervical pessary
  Arms: Cervical pessary

SUMMARY:
Preterm birth (PTB), defined as birth between 20 and 36 6/7 weeks, is responsible for the majority of the neonatal morbidity and mortality in the United States, and 35% of all U.S. healthcare spending on infants. Globally, about 28% of the 4 million annual neonatal deaths are directly attributable to PTB.

Preterm labor (PTL) is the final pathway for about 50% of all PTB. Tocolytic agents are drugs that can slow or stop labor contractions in the attempt to delay births preceded by PTL. Primary tocolysis is defined as tocolysis given on initial presentation of women with PTL. In most of these women, PTL stops, but as their risk of PTB remains high, some have advocated use of maintenance tocolysis, i.e. tocolysis after arrested PTL. So far, no maintenance tocolytic agent has been shown to be beneficial in preventing PTB.

The aim of this study is to evaluate the efficacy of maintenance tocolysis with Arabin pessary compared to standard care in singleton gestations with arrested PTL and with short transvaginal ultrasound (TVU) cervical length (CL) <25mm

ELIGIBILITY:
Inclusion Criteria:

* 18-50 ages
* Singleton pregnancy
* 24(0) - 34(6) weeks of gestation
* Arrested preterm labor after primary tocolysis
* Transvaginal ultrasound cervical length less than 25mm at admission
* Agreement to regular follow-up and provision of written informed consent

Exclusion Criteria:

* pessary and no cerclage in situ
* vaginal bleeding
* placeta previa/accreta
* multiple gestations
* <24(0) or >24(6) weeks of gestation
* Cervical dilatation greater than 3 cm
* Chorioamnionitis
* Major fetal abnormalities
* Abruptio placentae
* PPROM
* Polyhydramnios or oligohydramnios
* IUGR/FGR with or without Doppler abnormalities
* Preeclampsia or pregnancy-related hypertension

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Spontaneous preterm birth (SPTB) | Less than 34 weeks gestation

SECONDARY OUTCOMES:
Spontaneous preterm birth (SPTB) | Less than 37,35,32,28 and 24 weeks gestation
Gestational age at delivery | Delivery (at birth)
  mean gestational age at delivery
Latency | Delivery (at birth)
  mean latency in days (from randomization to delivery)
Birth weight | Delivery (at birth)
  mean birth weight in grams
Admission to neonatal intensive care unit | Delivery (at birth)
respiratory distress syndrome | Delivery (at birth)
low birth weight | Delivery (at birth)
  birth weight <2500 grams
intraventricular hemorrhage | Between birth and 28 days of age
  grade 3 or 4
neonatal mortality | Between birth and 28 days of age
  death of a live-born baby within the first 28 days of life

CONTACTS AND LOCATIONS:
Locations (1):
- University of Naples Federico II, Naples, Italy